CLINICAL TRIAL: NCT06123312
Title: Tri-modality Sampling Using Radial Probe Endobronchial Ultrasound for the Diagnosis of Peripheral Pulmonary Lesions- A Prospective Observational Pilot Study
Brief Title: Tri-modality Sampling Using Radial Probe Endobronchial Ultrasound for the Diagnosis of Peripheral Pulmonary Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Collaborators: Erbe-med (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2310-020-132
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lung Nodule
Keywords: Radial Probe Endobronchial Ultrasound; Pulmonary Nodule; Forceps Biopsy; Needle Aspiration; Cryobiopsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single intervention arm: Tri-modality biopsy (Experimental): Patients enrolled in this single arm will have lung nodules biopsied by Tri-modality (forceps biopsy, needle aspiration, and cryobiopsy)
  Interventions: Diagnostic Test: Tri-modality biopsy

INTERVENTIONS:
Diagnostic Test: Tri-modality biopsy — When the lung nodule is visualized by ultrathin bronchoscope (3mm) with RP-EBUS, Tri-modality biopsy is performed.

SUMMARY:
As the former radial probe endobronchial ultrasound (RP-EBUS) guided transbronchial forceps biopsy of peripheral pulmonary nodules has some limitations, the purpose of this study is to investigate a novel biopsy technique that combines forceps biopsy, needle aspiration, and transbronchial cryobiopsy in patients with peripheral pulmonary nodules.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label trial designed to assess the diagnostic accuracy and safety of the Tri-modality (forceps biopsy, needle aspiration, and transbronchial cryobiopsy) biopsy in patients with peripheral pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

* Patient with peripheral lung nodule less than 30mm on CT scan referred for biopsy
* Age ≥ 18
* Written informed consent after participant's information

Exclusion Criteria:

* Central lesion (visible on bronchoscope) or presence of metastatic lymph node (not requiring radial EBUS)
* Pure GGO lesion
* Patients at increased risk of bleeding

  1. Cannot stop agents such as antiplatelet agent or anticoagulant therapy
  2. Coagulopathy: Thrombocytopenia (< 100,000/mm3) or prolonged PT (INR > 1.5)
* Patient with existing or risk of pulmonary and cardiovascular decompensation
* Intolerance to sedation
* Vulnerable groups such as pregnant woman, breast feeding, etc.
* Previously diagnosed cancer patient who needs re-biopsy for genetic susceptibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield based on pathologic diagnosis | Time Frame: up to 6 months
  Diagnostic yield based on pathologic diagnosis is defined as percentage of definitive pathological diagnosis by transbronchial Tri-modality biopsy. If the bronchoscopic procedure fails to diagnose malignancy, the gold standard will be the results of additional procedures such as repeated bronchoscopic biopsy, percutaneous needle aspiration, surgical biopsy, or CT follow-up without any invasive procedure.

SECONDARY OUTCOMES:
Diagnostic yield based on clinical diagnosis | Time Frame: up to 6 months
  Diagnostic yield based on clinical diagnosis is defined as percentage of pathological diagnosis with suspicious results by transbronchial Tri-modality biopsy. If the bronchoscopic procedure fails to diagnose malignancy, the gold standard will be the results of additional procedures such as repeated bronchoscopic biopsy, percutaneous needle aspiration, surgical biopsy, or CT follow-up without any invasive procedure.
Adverse events | Time Frame: up to 1 week
  Occurrence of bleeding, pneumothorax, and infection events (during the procedure and within 1 week after the intervention). Bleeding will be assessed as the following scale (a. mild = self-limiting bleeding, manageable with suction alone and without the need for any specific intervention; b. moderate = use of any additional intervention such as instillation of ice-cold saline or vasoconstrictive drugs, or transient balloon tamponade, ; c. severe = additional prolonged monitoring or intensive care therapy after the procedure or if the bleeding was fatal). Pneumothorax will be assessed as the following scale (a. pneumothorax not requiring chest tube insertion; b. pneumothorax requiring chest tube insertion).

OTHER OUTCOMES:
Radial endobronchial ultrasound probe orientation | Time Frame: up to 1 day
  Lesion orientation regarding radial endobronchial ultrasound probe is assessed as the following scale (a. within, concentric; b. within, eccentric; c. adjacent; d. invisible).
Procedure time in minutes and seconds | Time Frame: up to 1 day
  The time spent in procedure begins with the insertion of bronchoscope into vocal cord and ends with removal of bronchoscope from vocal cord.
Diameter of cryoprobe | Time Frame: up to 1 day
  Diameter of cryoprobe use is assessed as the following scale (a. 1.1mm; b. 1.7mm).
Number of forceps biopsy | Time Frame: up to 1 day
  The number of forceps biopsy samples is assessed.
Number of needle aspiration | Time Frame: up to 1 day
  The number of needle aspiration samples is assessed.
Freezing time of cryoprobe in seconds | Time Frame: up to 1 day
  The freezing time of cryoprobe for sampling the lesions is assessed in seconds.
Biopsy size in millimeter | Time Frame: up to 1 month
  Size of biopsy tissue is assessed by pathologist for maximum and minimum diameter in millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Seop Eom, MD, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No